CLINICAL TRIAL: NCT02665234
Title: A Safety and Efficacy Study of Tavilermide Ophthalmic Solution for the Treatment of Dry Eye Disease
Brief Title: A Safety and Efficacy Study of Tavilermide (MIM-D3) Ophthalmic Solution for the Treatment of Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mimetogen Pharmaceuticals USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MIM-726
Record Dates: First submitted 2016-01-20; First posted 2016-01-27 (Estimated); Last update posted 2019-08-16 (Actual); Status verified 2019-08

CONDITIONS: Keratoconjunctivitis Sicca
Keywords: Dry Eye
MeSH Terms: conditions — Keratoconjunctivitis Sicca; Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Tavilermide Ophthalmic Solution (Active Comparator): 1% Tavilermide Ophthalmic Solution
  Interventions: Drug: 1% Tavilermide Ophthalmic Solution
- Vehicle Ophthalmic Solution (Placebo Comparator): Placebo Ophthalmic Solution
  Interventions: Drug: Placebo Ophthalmic Solution

INTERVENTIONS:
Drug: 1% Tavilermide Ophthalmic Solution — 1% Tavilermide BID Dosing
  Arms: Tavilermide Ophthalmic Solution
Drug: Placebo Ophthalmic Solution — Vehicle Ophthalmic Solution
  Arms: Vehicle Ophthalmic Solution

SUMMARY:
The purpose of this study is to assess the safety and efficacy of Tavilermide Ophthalmic Solution compared with Placebo Ophthalmic Solution in treating the signs and symptoms of dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Be at least 18 years of age.
* Provided written informed consent.
* Have a reported history of dry eye Have a history of use or desire to use eye drops for dry eye

Exclusion Criteria:

* Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal) at Visit 1.
* Be diagnosed with ocular rosacea, or any viral or bacterial disease of the cornea or conjunctiva, within the last 12 months.
* Have any planned ocular and/or lid surgeries over the study period.
* Have corrected visual acuity greater than or equal to +0.7 as assessed by Early Treatment of Diabetic Retinopathy Study (ETDRS) scale in both eyes at Visit .
* Have an uncontrolled systemic disease.
* Be a woman who is pregnant, nursing or planning a pregnancy.
* Be a woman of childbearing potential who is not using an acceptable means of birth control
* Have a known allergy and/or sensitivity to the test article or its components.
* Have a condition or be in a situation which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study
* Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 45 days of Visit 1 Be unable or unwilling to follow instructions, including participation in all study assessments and visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2016-01; Primary Completion 2017-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Total Corneal Fluorescein Staining Using The Ora Calibra Scale | Day 57
  An assessment of the total corneal fluorescein staining using the Ora Calibra Scale both immediately prior to and immediately following exposure to a challenge in a controlled adverse environment (CAE)
Ocular Discomfort Using The Ora Calibra Scale | Day 57
  A patient-reported subjective assessment of ocular discomfort recorded at each of the 5 office visits throughout the treatment period

SECONDARY OUTCOMES:
Total Corneal Fluorescein Staining Using The Ora Calibra Scale | Day 15
  An assessment of the total corneal fluorescein staining using the Ora Calibra Scale both immediately prior to and immediately following exposure to a challenge in a controlled adverse environment (CAE)
Ocular Surface Disease Index | Day 57
Ocular Dryness Using The Ora Calibra Scale | 8 weeks
  A patient-reported subjective assessment of ocular dryness recorded twice daily over the complete treatment period.

CONTACTS AND LOCATIONS:
Overall Officials: Garth Cumberlidge, PhD, Study Director — Mimetogen Pharmaceuticals USA, Inc.
Locations (1):
- MIM-726 Investigational Site, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No